CLINICAL TRIAL: NCT04859998
Title: Effects of Animal-assisted Therapy on the Physical Function and Communication of Adults With Autism: a Controlled Trial.
Brief Title: Effects of Animal-assisted Therapy on the Physical Function and Communication of Adults With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daniel Collado-Mateo (Other)
Collaborators: Asociación de Padres de Personas Con Autismo (APNA) (Unknown); Asociación Nuevo Horizonte (Unknown); Federación Autismo Madrid (Unknown)
Responsible Party: Sponsor-Investigator, Daniel Collado-Mateo, Assistant Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AATinAutism
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: dog-assisted; gait; postural; communication; Human-animal interaction; fall risk
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication; Human-Animal Interaction | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Two groups: one control (adults with autism that continues with their daily living and therapies) and one experimental group (adults with autism that receive the intervention program added to their daily living and therapies).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in this group will simply continue with their daily living and therapies. They will be assessed before and after the 10 week program but will not take part in it.
- Experimental group (Experimental): Participants in this group will take part in the 20 session dog-assisted therapy. This therapy will be added to their usual daily living and therapies. They will be assessed before and after the 10 week program.
  Interventions: Behavioral: dog-assisted therapy

INTERVENTIONS:
Behavioral: dog-assisted therapy — It will consist of 20 sessions conducted twice a week in the facilities of the association. It will involve different activities and physical exercises facilitated by the dogs. The program will be conducted in two associations (12 participants in each one, 6 belonging to the experimental and 6 belonging to the control group in each association) and in groups of three participants.
  Other Names: animal-assisted therapy; animal-assisted intervention
  Arms: Experimental group

SUMMARY:
The aim is to evaluate the effects of a dog-assisted therapy program on physical function and communication in a sample comprised of 24 adults with autism spectrum disorder. The sample will be divided into 2 groups, a control group and an experimental group. Changes after 10 weeks (20 sessions) will be compared between-groups.

DETAILED DESCRIPTION:
The intervention program will consist of 20 sessions conducted twice a week in the facilities of the collaborator associations. Each session will be conducted in groups of 3 participants and will last 30 minutes. It will include a welcome part, a main part (based on different activities and physical exercises with the dog) and a closing part to say goodbye to the dogs.

Physical function measures will be conducted before and after the completion of the study. The interaction and communication will be assessed during the sessions in the first, tenth and last ones.

ELIGIBILITY:
Inclusion Criteria:

* Older than 40 years
* With autism spectrum disorder
* Able to walk autonomously, without help from other people.
* Able to climb and descent stairs autonomously, without help from other people.

Exclusion Criteria:

* Medical condition that contraindicates the proximity or contact with the animals with the animals on the part of the user.
* Allergy to dog epithelium.
* Phobias to dogs.
* History of aggression to animals.
* Users who do not submit a signed informed consent form.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Changes in walking performance (10m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the ability to walk 10 meters in a corridor (time spent)
Changes in walking performance (6m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the ability to walk 6 meters in a corridor (time spent)

SECONDARY OUTCOMES:
Changes in balance and risk of falling | At baseline and inmediately after the intervention (within 7 days after the last session)
  Using the Tinetti Assessment Tool. Minimum score = 0. Maximum score for gait = 12 points; Maximum score for balance component = 16 points. Maximum total score = 28 points. Higher scores mean lower risk of falling.
Changes in communication without dog | At baseline and inmediately after the intervention (within 7 days after the last session)
  An observation scale designed by the group to evaluate the interaction and communication with other people. It is comprised by 14 items, scored as 1 (yes) and 0 (no). Minimum score = 0; Maximum score = 14. Higher scores mean higher communication.
Changes in communication with dog | During sessions (first, intermediate and last one)
  An observation scale designed by the group to evaluate the interaction and communication with the dogs and other people. It is comprised by 38 items, scored as 1 (yes) and 0 (no). Minimum score = 0; Maximum score = 38. Higher scores mean higher communication.
Changes in the ability to climb and descend stairs | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the ability to climb and descend stairs (10 steps)
Changes in step length (6m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the step length walking 6 meters in a corridor
Changes in step length (10m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the step length walking 10 meters in a corridor
Changes in cadence (6m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the cadence walking 6 meters in a corridor
Changes in cadence (10m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the cadence walking 10 meters in a corridor
Changes in duration of phases in the gait cycle (6m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the duration of phases in the gait cycle walking 6 meters in a corridor
Changes in duration of phases in the gait cycle (10m) | At baseline and inmediately after the intervention (within 7 days after the last session)
  Evaluation of the duration of phases in the gait cycle walking 10 meters in a corridor

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Collado-Mateo, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- King Juan Carlos University, Móstoles, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No